CLINICAL TRIAL: NCT01204190
Title: Multicenter, Open-label, Randomized Study to Evaluate Inhibition of Ovulation During Treatment With Three Transdermal Patch Formulations Containing 0.55 mg Ethinylestradiol (EE) and 2.10 mg Gestodene (GSD) or 0.35 mg EE and 0.67 mg GSD or 0.275 mg EE and 1.05 mg GSD in Healthy Young Female Volunteers Over a Period of 3 Treatment Cycles
Brief Title: Investigation of Three Contraceptive Hormone Patches in Regard to Inhibition of Ovulation Following Application Over 3 Treatment Cycles in Healthy, Young Women.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15264; 2010-021255-81 (EudraCT Number)
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Contraception
Keywords: Administration; Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Gestodene/EE Patch (BAY86-5016)
- Arm 2 (Experimental)
  Interventions: Drug: Gestodene/EE Patch (BAY86-5016)
- Arm 3 (Experimental)
  Interventions: Drug: Gestodene/EE Patch (BAY86-5016)

INTERVENTIONS:
Drug: Gestodene/EE Patch (BAY86-5016) — 0.55 mg ethinyl estradiol (EE) + 2.1 mg gestodene (GSD) per patch; 3 treatment cycles; 21 days per treatment cycle, i.e. 3 x 7 days patch-wearing phase and a patch-free interval of 7 days
  Arms: Arm 1
Drug: Gestodene/EE Patch (BAY86-5016) — 0.35 mg ethinyl estradiol (EE) + 0.67 mg gestodene (GSD) per patch; 3 treatment cycles; 21 days per treatment cycle, i.e. 3 x 7 days patch-wearing phase and a patch-free interval of 7 days
  Arms: Arm 2
Drug: Gestodene/EE Patch (BAY86-5016) — 0.275 mg ethiny estradiol (EE) + 1.05 mg gestodene (GSD) per patch; 3 treatment cycles; 21 days per treatment cycle, i.e. 3 x 7 days patch-wearing phase and a patch-free interval of 7 days
  Arms: Arm 3

SUMMARY:
The primary objective of this trial is to examine whether ovulation is suppressed after use of hormone patches containing different dosages of ethinyl estradiol (EE) and gestodene (GSD) for 3 treatment cycles. To this end, the blood levels of endogenous hormones (hormones produced by your body) will be measured and transvaginal ultrasound examinations will be conducted at regular intervals. In addition, the concentrations of the administered hormones EE and GSD in blood will be determined in regular intervals.

With regard to the tolerability of the hormone patches subjects will be asked regularly how they feel and blood pressure, pulse and body weight will be determined. In addition, blood and urine safety examinations will be conducted at defined timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers
* age 18 - 35 years (smoker not older than 30 years, inclusive)
* ovulatory pre-treatment cycle

Exclusion Criteria:

* Contraindications for use of combined (estrogen/gestodene) contraceptive (e.g. history of venous or arterial thromboembolic disease)
* Regular intake of medication other than Oral Contraception
* Clinically relevant findings (blood pressure, physical and gynecological examination, laboratory examination)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Hoogland score to evaluate the inhibition of ovulation | After 2 months

SECONDARY OUTCOMES:
Blood level time course of gonadotropins i.e. follicle stimulating hormone (FSH) and luteinizing formone (LH) as well as steroid hormones estradiol and progesterone | After 2 months
Follicle size measured by transvaginal ultrasound examination | After 2 months
Pharmacokinetics of ethinyl estradiol (EE), gestodene (GSD) and sex hormone binding globuline (SHBG) | After 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Berlin, State of Berlin, Germany
- Groningen, Netherlands

REFERENCES:
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu